## UNIVERSITY OF CALIFORNIA, SAN DIEGO

UCSD

BERKELEY • DAVIS • IRVINE • LOS ANGELES • MERCED • RIVERSIDE • SAN DIEGO • SAN FRANCISCO



OFFICE OF:

gfeld@ucsd.edu

GREGORY K. FELD, M.D

PROFESSOR OF MEDICINE DIRECTOR EP PROGRAM

9444 MEDICAL CENTER DR MC 7411 LA JOLLA, CALIFORNIA 92037

SANTA BARBARA • SANTA CRUZ

DIVISION OF CARDIOVASCULAR MEDICINE TELEPHONE: (858) 657-8530 NIGHTS & WEEKENDS: (619) 543-6737

FAX: (858) 657-5054

Date: November 15, 2024

To: Whom it may Concern

Re: Project # 130663

NCT02154750

Evaluation of AV Delay Optimization vs. Intrinsic Conduction in Patients with Long PR Intervals

Receiving Dual Chamber Pacemakers for Symptomatic Bradycardia.

Statistical Analysis Variables are displayed as the mean  $\pm$  1SD. Categorical variables are presented as number and percentage. For comparisons of the baseline categorical variable between groups, chi-square test was used. Wilcoxon signed-rank test was used to compare each variable between baseline and 6 months after randomization. The change in each parameter was compared between each group using the Mann-Whitney U test. A p value of < 0.05 was considered statistical significance. Analyses were performed using SPSS version 23 (IBM corporation, Chicago, Illinois).

If there are any questions or concerns regarding this submission, please contact Benyraemon Batenga, Research Coordinator, at 858-246-2405. Thank you for your consideration in this matter.

Sincerely,

Gregory Feld, MD /bb Professor of Medicine

Director Cardiac Electrophysiology Program

University of California, San Diego